CLINICAL TRIAL: NCT01805726
Title: Success of Sedation During Bronchoscopy: Comparison of the Effects of Dexmedetomidine, Alfentanil and Local Anesthesia
Brief Title: Sedation During Bronchoscopy:Dexmedetomidine vs Alfentanil
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Saint-Joseph University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FM235
Record Dates: First submitted 2013-02-17; First posted 2013-03-06 (Estimated); Last update posted 2014-11-25 (Estimated); Status verified 2014-11

CONDITIONS: Bronchoscopy; Conscious Sedation
Keywords: bronchoscopy; sedation; pulmonary function; tolerance; xylocain; dexmedetomidine; alfentanil
MeSH Terms: interventions — Alfentanil; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Xylocain (C) (Placebo Comparator): (C): Local anesthesia
  Interventions: Drug: xylocain
- Alfentanil Group + Xylocain (A) (Active Comparator): Local anesthesia and Alfentanil
  Interventions: Drug: Alfentanil
- Dexmedetomidine Group + Xylocain (D) (Active Comparator): Local anesthesia and dexmedetomidine
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: xylocain — Xylocain: (C): Local anesthesia 1% 25 ml in total (bronchoscopy) + saline serum
  Other Names: Xylocain only
  Arms: Xylocain (C)
Drug: Alfentanil — (A) Local anesthesia 1% 25 ml in total (bronchoscopy) + saline serum (slow perfusion for 10 minutes) + alfentanil 10 mcg / kg (slow injection in 5 seconds)
  Other Names: Alfentanil as morphinics short acting
  Arms: Alfentanil Group + Xylocain (A)
Drug: Dexmedetomidine — (D) Local anesthesia 1% 25 ml in total (bronchoscopy) + dexmedetomidine 0.5 mcg / kg (slow perfusion for 10 minutes) + 2 ml saline (slow injection for 5 seconds)
  Other Names: Dexmedetomidine as awake sedation
  Arms: Dexmedetomidine Group + Xylocain (D)

SUMMARY:
The purpose of this study is to find the best sedation necessary for patients undergoing bronchoscopy. Patients are randomized to three different regimes of sedation during bronchoscopy were studied:

1. - Group standard/control: local anesthesia only(C)
2. - Group alfentanil + local anesthesia(A)
3. - Group dexmedetomidine + local anesthesia(D) The primary endpoint is the bronchoscopy score. Secondary endpoints are: Level of sedation and tolerance bronchoscopy examination. Measured parameters on the safety of examination are: the lowest saturation, needs to supplemental oxygen, amnesia , choking sensation or chest pain and if the patient is ready or not to undertake bronchoscopy second time in his life if necessary. Endtidal CO2, Respiratory rate, Blood pressure, Heart rate, level of oxygen are collected every 5 minutes before, during and after the bronchoscopy.

DETAILED DESCRIPTION:
BACKGROUND:

1. Problem:

   The endoscopy of the tracheobronchial tree by endoscopy is an act very common in the daily activity of pulmonologists. The indications for bronchoscopy are multiple and include infectious causes, tumor, systemic disease, foreign bodies and other indications. It can be diagnostic or therapeutic purposes. Bronchoscopy is an invasive but rarely, however, induced severe complications (respiratory failure, hemodynamic collapse, massive bleeding ...). However, tolerance to the examination varies significantly between patients [1-3]. Different signs and symptoms include desaturation, chest pain, choking sensation and cough. These effects are likely to alter patient comfort during the procedure and the quality of it. To further improve the tolerance operators have resorted to various techniques. A first step in improving the comfort is a good local anesthesia using spray or swab intra nasal base and lidocaine anesthesia of the airway (trachea, carina and bronchi) during the examination. The second step involves the use of intravenous sedation [1, 3-14].
2. Background:

Until now, there is no standardized protocol for the best product and the best dose to use for sedation of patients. Several studies have been done comparing different drug or drug combination in the benzodiazepine family, ketamine or morphine with varying results and not leading in most cases to allow conclusions to establish clear guidelines regarding the use or no sedation plus local anesthesia and sedation dose of this [1, 3, 5, 8, 15]. Especially, for fear of adverse effects of sedation on respiratory function, many pulmonologists far are a little hesitant about the administration of sedatives during bronchoscopy. Dexmedetomidine is a new molecule sedation which is approved for its sedative effect while holding a revival meeting described as "awake sedation." [12, 16-22]

DESCRIPTION:

The aim of this randomized controlled trial was to evaluate the feasibility and safety of three different regimes of sedation during bronchoscopy:

* Group standard / control (local anesthesia only): (C)
* Group alfentanil (+ local anesthesia): (A)
* Group dexmedetomidine (+ local anesthesia): (D)

The primary endpoint is:

1. / Feasibility / tolerance of bronchoscopy by the "score bronchoscopy" which includes:

   * The movement of the vocal cords (4 levels)
   * Cough (4 levels)
   * Movement members (4 levels)

   Secondary objectives:
2. / level sedation for bronchoscopy:

   * Level of sedation achieved according to the objective using: Nursing Instrument for the Communication of Sedation (NICS) (7 levels).
   * Dose of midazolam necessary complementary in each group. Midazolam to give to the judgment of the operator (if necessary) is predetermined speed (1 mg each minute) to the level of sedation (-1) "Level of sedation achieved according to the objective using: Nursing Instrument for the communication of Sedation (NICS)".
3. / Tolerance examination:

   * During the procedure
   * At the end of the procedure
   * After 1 hour of the end of the examination

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted for diagnostic flexible bronchoscopy in the endoscopy department

Exclusion Criteria:

* Bronchoscopy outside the endoscopy unit
* Tracheal stenosis
* SpO2 <90% in the open air
* Bradycardia <55 per minute
* Atrioventricular block
* Heart failure known (EF <40%)
* Alcoholism (> 5 drinks per week)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2013-02; Primary Completion 2013-03 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Bronchoscopy score | At the end of the bronchoscopy procedure
  Feasibility / tolerance of bronchoscopy by the "score bronchoscopy" which includes:
  * The movement of the vocal cords (4 levels)
  * Cough (4 levels)
  * Movement members (4 levels) Scale will be between: minimum 3 and maximum 16

SECONDARY OUTCOMES:
Level of sedation for bronchoscopy | At the end of the bronchoscopy procedure
  * Level of sedation achieved according to the objective using: Nursing Instrument for the Communication of Sedation (NICS) (7 levels).
  * Dose of midazolam necessary complementary in each group. Dormicum to give to the judgment of the operator (if necessary) is predetermined speed (1 mg each minute) to the level of sedation (-1) "Level of sedation achieved according to the objective using: Nursing Instrument for the communication of Sedation (NICS) "

OTHER OUTCOMES:
Tolerance of examination | During, at the end and one hour after the bronchoscopy.
  Visual Analogic Scale from 0-10 to evaluate the tolerance of the procedure:
  * During the procedure
  * At the end of the procedure
  * After 1 hour of the end of the examination

CONTACTS AND LOCATIONS:
Overall Officials: Moussa A Riachy, MD, FCCP, Principal Investigator — Saint-Joseph University
Locations (1):
- Hotel Dieu de France Hospital, Beirut, Lebanon